CLINICAL TRIAL: NCT06934759
Title: Impact and Lived Experience of Parents of a Child With a Large or Giant Congenital Melanocytic Nevus (PANGEA Study) : A National Qualitative Study
Brief Title: Impact and Lived Experience of Parents of a Child With a Large or Giant Congenital Melanocytic Nevus
Acronym: PANGEA
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); Hôpital Necker-Enfants Malades (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Brest (Other); Annecy Hospital, France (Unknown); Centre Hospitalier Universitaire Dijon (Other); Nantes University Hospital (Other); University Hospital, Grenoble (Other); Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Principal Investigator, Anne Claire BURSZTEJN, Clinical Professor and Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI238
Record Dates: First submitted 2025-04-06; First posted 2025-04-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Congenital Melanocytic Nevi; Congenital Melanocytic Nevus; Parent; Psychology, Social
Keywords: parents; congenital melanocytic nevus; congenital melanocytic nevi; psychology; lived experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with congenital melanocytic nevus
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — There is no intervention

SUMMARY:
The goal of this observational study is to describe the experiences of parents at the birth of a child with a large or giant congenital melanocytic nevus through semi-structured interviews, and to identify potential intervention strategies to improve their care and support.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Willing to participate in a semi-structured interview
* Has received full information about the research and has not objected to participating or to the use of their data
* Able to understand and speak French
* Parent of a child under 18 years of age

Exclusion Criteria:

* Under 18 years of age
* Not willing to participate
* Currently under legal protection (e.g., guardianship or curatorship)
* Cognitive and/or psychological impairments preventing participation in a semi-structured interview
* Poor understanding and/or expression of the French language
* Parent of a child over 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include parents of children with a large or giant congenital melanocytic nevus who are being followed at the university hospitals (CHRU) of Nancy, Marseille, Nantes, Dijon, Necker, Nice, Brest, Annecy, Grenoble and Saint Pierre.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Results of the Semi-Structured Interviews with Parents | Socio-demographic data and interview transcripts will be collected during the semi-structured interviews (lasting between 30 minutes and 1 hour), thus at a single time point (Day 1). No follow-up is required.
  Analysis of the interview transcripts = verbatim analysis Individual semi-structured interviews will be conducted via videoconference, with an estimated duration of 30 minutes to 1 hour. An interview guide has been developed to define the key dimensions to be explored. Each interview will be audio-recorded using a voice recorder and then fully transcribed.
  The interviews will undergo a thematic content analysis to identify meaningful patterns ("nodes of meaning") within participants' narratives, using an inductive approach. A double coding will be performed by two investigators on five interviews to strengthen the thematic framework. The remaining interviews will be coded by a single investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France, France

IPD SHARING:
Plan to Share IPD: Undecided